CLINICAL TRIAL: NCT03451903
Title: Which Factors Influence the Duration and the Success of Mechanical Thrombectomy During the Acute Phase of Cerebral Infarction?
Acronym: REPAIR-FC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2017/348
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-02

CONDITIONS: Acute Stroke
Keywords: stroke; thrombectomy; procedure time; revascularisation; thrombolytic therapy
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mechanical thrombectomy group: Patients with acute stroke treated by mechanical thrombectomy.
  Interventions: Procedure: Mechanical thrombectomy
- Combined procedure group: Patients with acute stroke treated by intravenous thrombolysis (with actilyse) and mechanical thrombectomy.
  Interventions: Drug: Actilyse; Procedure: Mechanical thrombectomy

INTERVENTIONS:
Drug: Actilyse — Actilyse is the intra-venous agent used for intra-venous thrombolysis in the acute phase of cerebral infarction.
  Other Names: rtPA
  Groups: Combined procedure group
Procedure: Mechanical thrombectomy — Mechanical thrombectomy is an endovascular procedure by which an arterial clot is retrieved, in order to reperfuse the brain.

SUMMARY:
This study aims to identify factors influencing the time span and success of reperfusion after a mechanical thrombectomy in the acute phase of cerebral infarction, and in particular the effect of intra-venous thrombolysis.

DETAILED DESCRIPTION:
Mechanical thrombectomy (MT), associated with standard IV thrombolysis (IVT) treatment, is effective during the acute phase of cerebral infarction with proximal occlusion of the anterior circulation in reducing disability at three months. MT-only treatment has only been assessed retrospectively in subgroups of controlled studies, with a significant difference in favour of the treatment. These results have led to a discussion about the benefits of MT without IVT in cases of proximal occlusion or carotid terminus occlusion. Recent data are in favour of a better prognosis for patients benefiting from a combined procedure. The impact of IVT on the implementation of MT is widely disputed, in particular the speed of execution, which could be enhanced by IVT. The factors influencing the time span and success of reperfusion after an MT are still not well-known, IVT in particular. The investigators have made the assumption that IVT could have an effect on the success of MT by shortening the duration of the procedure and increasing the likelihood of satisfactory revascularisation.

The investigators carried out a retrospective study based on data gathered prospectively by the Franche-Comté Stroke Registry. The investigators also considered other factors which could have affected the duration of the procedure or the rate of satisfactory revascularisation, including location of infarct, thrombus size and stroke aetiology.

Hypothesis: the investigators have made the assumption that IVT could have an effect on the success of MT by shortening the duration of the procedure and increasing the likelihood of satisfactory revascularisation.

ELIGIBILITY:
Inclusion Criteria:

* acute phase of cerebral infarction
* all patients who had undergone an arteriography for cerebral infarction prior to mechanical thrombectomy at CHRU Besançon
* from 1st January 2015 to 31st December 2016

Exclusion Criteria:

* Patients whose procedures were interrupted (puncture failure, catheterisation of the common or internal carotid artery failure)
* Patients whose arteries were recanalised during the diagnostic arteriography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had undergone an arteriography for cerebral infarction prior to mechanical thrombectomy at CHRU Besançon. Data are prospectively collected in the Franche-Comté Stroke Registry.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Duration of the procedure | From the beginning of mechanical thrombectomy to the end of the procedure.
  It is the period of time between when the artery is punctured and when the first image from the first cerebral angiographic test is acquired after revascularisation, which is used to calculate the rate of revascularisation.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Bonnet, MD, Principal Investigator — J Minjoz Besancon university Hospital

IPD SHARING:
Plan to Share IPD: No